CLINICAL TRIAL: NCT06494800
Title: Added Value of 18F-FDG PET/CT in Lung Cancer
Brief Title: Added Value of PET/CT in Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mennatallah Ahmed Ragheb, resident, nuclear and oncology medicine department, Sohag university, Sohag University
Other Study IDs: PET/CT in lung cancer
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
Keywords: PET-CT; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pathologically proved lung cancer patient: All the pathologically proved lung cancer patients by true cut needle biobsy are enrolled in the study.
  the true cute needle biobsy procedure performed by two interventional radiologists and a pathologist. TCNB was guided by the use of a 16-detector CT device after local anesthesia is done and done either by ultrasound guidance or CT guidance.
  Interventions: Diagnostic Test: True cut needle biobsy

INTERVENTIONS:
Diagnostic Test: True cut needle biobsy — The biobsy procedure done at the radiology department and the cores are examined by the pathology department, the patient lie prone, supine or in lateral decubitus according to the location of the lesion. A thoracic CT scan was performed first to evaluate the needle pathway and distance from the puncture site to the lesion. The needle pathway was selected to avoid bone, visible vessels, bullae, and fissures. The puncture site was chosen by the CT gantry laser lights and landmarks using a homemade radiopaque grid on the patient's skin. Local anaesthesia was induced with 5 mL of 2% lidocaine. An 18-G coaxial needle was used to puncture the lung, and a repeat CT scan was performed to evaluate the site of the needle. When the needle tip reached the lesion, the specimen was obtained by pressing the trigger of the needle. The specimen was reviewed by the pathologist.The specimen was placed in 10% formaldehyde for pathological examination.
  Other Names: TCNB

SUMMARY:
Assess the value of PET/CT in the diagnosis, staging, response evaluation, and relapse monitoring of lung cancer.

DETAILED DESCRIPTION:
Lung cancer is a leading cause of cancer-related mortality worldwide, accounted for 1.80 million deaths in 2020.(1)Egyptian statistics showed that lung cancer in men represents 8.2% of among all cancers of men according to the Egyptian National Cancer Program in 2014 (3).Epidemiological data indicate that the main risk factor for the development of lung cancer is cigarette smoking.(4)Lung cancer is histologically divided into: Non-small-cell lung cancer (NSCLC), which accounts for 85% of cases and Small cell lung cancer (SCLC).(5)Due to absence of screening, most patients with lung cancer are not diagnosed until later stages, when the prognosis is poor.(6)Radiologic manifestations of bronchogenic carcinoma include obstructive pneumonitis or atelectasis, lung nodule or mass, apical mass, cavitated mass, or nodule or mass associated with lymphadenopathy(6)Conventional chest radiography, computed tomography (CT), magnetic resonance imaging, radionuclide scintigraphy, and positron emission tomography (PET) all have been used for NSCLC staging.(7)PET/CT is a well-established radiological modality with high diagnostic accuracy in metastases detection compared to usual CT. Also, it has been reported that up to 10% of patients with bronchogenic carcinoma are found to have metastases on PET/CT that were not detected on CT with subsequent different patients' staging. The high accuracy of PET/CT in tumor staging makes it important for the treatment strategy of either surgical treatment, radiotherapy, or chemotherapy. Also, it becomes essential during the follow-up to detect recurrence. PET/CT shows a higher ability to evaluate the early response to the treatment as chemotherapy by its ability to detect the metabolic response even before the size change.(8)The prognosis of lung tumors depends on early and accurate staging as well as the histopathological type of the primary tumor, with the squamous cell carcinoma type regarded to be of a worse prognosis than that of adenocarcinoma.(9)

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven lung cancer patients.

Exclusion Criteria:

* Patients with second malignancy.
* Severely ill patient (patient with disturbed consciousness level, or couldn't lie during the imaging).
* Uncontrolled diabetic patient with blood glucose level more than 200mg\dl.
* Pregnant women.
* Patient age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the pathologically proved lung cancer patient in the oncology department at the sohag oncology Centre.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of PET CT in diagnosis of lung cancer | 1 Year
  using the qualitative and quantitative measuring including the SUV max value in detection of the malignant potentiality of the pulmonary nodule or mass comparing it with the pathological result
Value of PET CT in staging of lung cancer | 1 Year
  using the PET CT in TNM staging with better detection of pleural , mediastinal extension /involvement, the value and accuracy of PET in detecting the potential malignancy of the mediastinal lymph nodes even the subcentemetric lymph nodes not adequately assessed by the usual CT.
predicting the pathological subtype of lung cancer using the morphological and PET CT of pathologically proved lung masses | 1 Year
  assessing the morphology of the lung mass including density, solid, subsolid and soft nodule.
  site of the nodule/mass peripheral or centrally located. presence of cavitation or cystic changes. presence of speculated or irregular margin. measuring the SUV max and comparing it with the pathology of each mass/nodule.
Differentiating between the primary mass and associated consolidation if present | 1 Year
  using the PET CT (mainly the qualitative assessment) in differentiating the primary mass from the associated consolidation-atelectasis around

SECONDARY OUTCOMES:
assessment of the pleural thickening/effusion associated with the primary mass | 1 Year
  assessing the qualitative and quantitative assessing the pleural thickening if found for differentiating the pleural involvement from the inflammatory pleural thickening
presence of enlarged axillary Lns | 1 Year
  assessing the activity of enlarged axillary Lns by measuring the SUV value
assessing the Vocal cord paralysis in the pan-coast tumor | 1 Year
  using the morphological assessment of the lower CT neck scans and the adduction of the vocal cord and the atrophic changes of the Muscle and loss of vocal cord physiological activity.

CONTACTS AND LOCATIONS:
Overall Officials: mai sayed khalifa, MD, Principal Investigator — lecturer; doaa ibrahim mohamed, MD, Principal Investigator — lecturer

REFERENCES:
- [Background] Archer JM, Truong MT, Shroff GS, Godoy MCB, Marom EM. Imaging of Lung Cancer Staging. Semin Respir Crit Care Med. 2022 Dec;43(6):862-873. doi: 10.1055/s-0042-1753476. Epub 2022 Jul 10. PMID 35815631
- [Background] Laguna JC, Garcia-Pardo M, Alessi J, Barrios C, Singh N, Al-Shamsi HO, Loong H, Ferriol M, Recondo G, Mezquita L. Geographic differences in lung cancer: focus on carcinogens, genetic predisposition, and molecular epidemiology. Ther Adv Med Oncol. 2024 Mar 6;16:17588359241231260. doi: 10.1177/17588359241231260. eCollection 2024. PMID 38455708
- [Background] Panunzio A, Sartori P. Lung Cancer and Radiological Imaging. Curr Radiopharm. 2020;13(3):238-242. doi: 10.2174/1874471013666200523161849. PMID 32445458
- [Background] Kandathil A, Subramaniam RM. FDG PET/CT for Primary Staging of Lung Cancer and Mesothelioma. Semin Nucl Med. 2022 Nov;52(6):650-661. doi: 10.1053/j.semnuclmed.2022.04.011. Epub 2022 Jun 20. PMID 35738910
- See also: Contrast computed tomography versus PET/CT in the assessment of bronchogenic carcinoma — https://doi.org/10.4103/epj.epj_49_18
- See also: Role of CT in differentiation between subtypes of lung cancer; is it possible? — https://doi.org/10.1186/s43168-020-00027-w
- See also: PET-CT in Lung Cancer — https://doi.org/10.1007/978-3-031-10090-1_5
- See also: FDG-PET/CT tumor to liver SUV ratio (TLR), tumor SUVmax, and tumor size: Can this help in differentiating squamous cell carcinoma from adenocarcinoma of the lung? — https://doi.org/10.1186/s43055-022-00782-4